CLINICAL TRIAL: NCT00925834
Title: Effects of Suggestive Components of Therapeutical Interventions on the Diameter of Coronary Arteries
Brief Title: Suggestive Effects on the Diameter of Coronary Arteries
Acronym: SUGO-KO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); German Heart Center (Other)
Responsible Party: Dr. Joram Ronel, Dr. Karin Meissner, Technische Universität München
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SUGOKO
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2009-06-22 (Estimated); Status verified 2009-06

CONDITIONS: Coronary Circulation
Keywords: Coronary angiography; Placebo effect; Suggestion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sodium chloride (Placebo Comparator): Control arm "A": Hidden intracoronary infusion of 5ml sodium chloride
  Interventions: Behavioral: Verbal suggestions
- Sodium chloride and verbal suggestions (Experimental): Experimental arm "A": Open intracoronary infusion of 5ml sodium chloride plus the suggestion of a vasodilatory effect on coronary vessels
  Interventions: Behavioral: Verbal suggestions
- Nitroglycerin (Active Comparator): Control arm "B": Hidden intracoronary infusion of 0.01mg nitroglycerin in 5 ml sodium chloride
  Interventions: Behavioral: Verbal suggestions
- Nitroglycerin and verbal suggestions (Experimental): Control arm "B": Open intracoronary infusion of 0.01 mg nitroglycerin in 5 ml sodium chloride plus the suggestion of a vasodilatory effect on cardiac vessels
  Interventions: Behavioral: Verbal suggestions

INTERVENTIONS:
Behavioral: Verbal suggestions — Verbal suggestions of a vasodilatory effect on cardiac vessels

SUMMARY:
The aim of this randomized controlled pilot study was to answer the following questions:

1. Is it possible to affect the diameter of coronary arteries through a placebo injection, which is administered intracoronarily together with a standardized verbal suggestion of coronary vasodilation?
2. Is it possible to affect the diameter of coronary arteries through a pharmacologically underdosed nitroglycerine injection, which is administered intracoronarily together with a standardized verbal suggestion of coronary vasodilation?

DETAILED DESCRIPTION:
The present study is a randomized controlled double-blind single center study in order to investigate the effects of verbal suggestions ('vasodilatation') in combination with either a placebo-intervention (sodium chloride 0.9%) or an underdosed vasodilating medication (nitroglycerine) on the diameter of coronary arteries. 60 patients with a clinical indication to undergo a coronary angiogram were recruited in the German Heart Centre Munich. Patients with acute myocardial events and the necessity for coronary intervention were excluded from the study. Patients were randomized into one of four arms of the two experiments:

Experiment A: Intracoronary (i.c.) placebo-infusion together with a standardized verbal suggestion of coronary vasodilation vs. i.c. placebo-infusion without verbal suggestion.

Experiment B: i.c. infusion of a very low dosed nitroglycerin together with a standardized verbal suggestion of coronary vasodilation vs. i.c. nitroglycerine infusion without verbal suggestion.

To our best knowledge this study is the first to investigate the modulating effects of verbal suggestions going along with medical interventions on the diameter of coronary arteries during heart catheterization.

ELIGIBILITY:
Inclusion Criteria:

* medical indication for heart catheterization
* written informed consent

Exclusion Criteria:

* acute myocardial infarction
* acute elevation of cardiac enzymes
* regular intake of drugs containing nitroglycerin
* intolerance of nitroglycerin
* hypotension
* renal insufficiency
* diabetes mellitus
* hyperthyroidism
* pregnancy
* acute psychiatric disease
* cognitive impairment
* prinzmetal's angina

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Stenosis Diameter (Quantitative Coronary Analysis) | 60 sec after intervention

SECONDARY OUTCOMES:
Heart rate | immediately before and after intervention
Systolic blood pressure | immediately before and after intervention
Diastolic blood pressure | immediately before and after intervention
Chest Pain | immediately before and after intervention
Subjective distress | immediately before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Joram Ronel, M.D., Principal Investigator — Technical University of Munich; Karin Meißner, M.D., Principal Investigator — Ludwig-Maximilians-Universität München; Julinda Mehilli, M.D., Principal Investigator — Deutsches Herzzentrum München
Locations (1):
- Department of Psychosomatic Medicine, Technische Universität München, Munich, Germany